CLINICAL TRIAL: NCT05313841
Title: Novel Equation for Estimating Intraperitoneal Pressure in Patients on Peritoneal Dialysis Patients
Brief Title: Novel Equation for Estimating Intraperitoneal Pressure
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Clinical Professor in Renal Division, Department of Medicine, Peking University First Hospital
Other Study IDs: IPP equation
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Intraperitoneal Pressure; Peritoneal Dialysis; Equation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intraperitoneal Pressure is associated with the complications of increased intra-abdominal pressure in peritoneal dialysis patients. Due to the complicated operations, routine measurement of hydrostatic intraperitoneal pressure is not used routinely in adult peritoneal dialysis patients. There ars some limitions in equations from previous studies, such as the sample size was small , and the study population was limited. In the study, we aim to develop and validate an equation for estimating intraperitoneal pressure in peritoneal patients.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis patients
* Dialysis length >1 month
* Aged 18-80 years
* Injection volume of peritoneal dialysis solution>1500ml

Exclusion Criteria:

* Acute complications （ peritonities, cardiovascular and cerebrovascular diseases) to hospitalization 1 month prior to the study
* History of abdominal surgery and trauma 1 month prior to the study
* Previous history of hernia, leakage, or thoracoabdominal fistula
* Can't come for a follow-up visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All peritoneal dialysis patients meet the inclusion and exclusion criteria in a single center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Novel equation development | July 17, 2021 to September 30, 2021
  Developed equation for estimating intraperitoneal pressure in peritoneal dialysis patients
Novel equation validation | October 1,2021 to October 31,2021
  Validate the novel equation with intraperitoneal pressure obtained by Durand method

CONTACTS AND LOCATIONS:
Locations (1):
- Jie Dong, Beijing, Beijing Municipality, China